CLINICAL TRIAL: NCT04928521
Title: Comparison of Postoperative Analgesic Efficacy of Erector Spinae Plane Block With 20 ml and 30 ml Bupivacaine Volumes in Cardiac Surgery
Brief Title: Erector Spinae Plane (ESP) Block With 20 ml Versus 30 ml in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Eda Balci, Principal investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MH2.3
Record Dates: First submitted 2021-06-06; First posted 2021-06-16 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Surgery; Postoperative Pain
Keywords: erector spinae plane block; local anesthetic volume; bupivacaine; sternotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block with 20 mL local anesthetic solution (Active Comparator): An erector spinae plane block will be performed at the level of the 5th thoracic vertebrae with 20 mL of 0.25% bupivacaine solution under ultrasound guidance before the operation.
  Interventions: Procedure: bilateral erector spinae plane block with 20 mL 0.25 % bupivacaine
- ESP block with 30 mL local anesthetic solution (Active Comparator): An erector spinae plane block will be performed at the level of the 5th thoracic vertebrae with 30 mL of 0.25% bupivacaine solution under ultrasound guidance before the operation.
  Interventions: Procedure: bilateral erector spinae plane block with 30 mL 0.25 % bupivacaine

INTERVENTIONS:
Procedure: bilateral erector spinae plane block with 30 mL 0.25 % bupivacaine — Preoperative, awake, bilateral, ultrasound-guided erector spinae plane block with 30 mL 0.25 % bupivacaine
  Other Names: 30 mL
  Arms: ESP block with 30 mL local anesthetic solution
Procedure: bilateral erector spinae plane block with 20 mL 0.25 % bupivacaine — Preoperative, awake, bilateral, ultrasound-guided erector spinae plane block with 20 mL 0.25 % bupivacaine
  Other Names: 20 mL
  Arms: ESP block with 20 mL local anesthetic solution

SUMMARY:
Even though erector spinae plane (ESP) block is shown to be efficient in cardiac surgery, it is still controversial how much volume is necessary for efficient analgesic effect for sternotomy and drain tube pain relief. This study aims to investigate the optimal local anesthetic volume (20 mL versus 30 mL) with ESP block for open-heart cardiac surgery.

DETAILED DESCRIPTION:
In cardiac surgery, the most common cause of pain during the first two days postoperatively is median sternotomy. In a study in which 705 patients who had undergone cardiac surgery were followed up prospectively, postoperative 24 hours pain scores ranging from 5.3 to 6.5 out of 10 with deep breathing and coughing were shown. In these patients, it may increase the frequency of atelectasis due to reasons such as failure in pain control, weak coughing, and limitation of movement, and these may lead increase in morbidity and hospital stay. Although nonsteroidal analgesics and opioids are used successfully in the control of this severe pain, they are far from being ideal analgesics alone due to their side effects such as kidney damage, bleeding risk, sedation, respiratory depression, itching, nausea, and vomiting. The complications of neuraxial techniques seem to be the disadvantages of these methods. Erector spinae plane (ESP) block is one of the regional anesthesia techniques that has been shown to be effective in reducing sternotomy pain in sternotomy-guided cardiac surgeries.

The Erector spinae plane (ESP) block was first described by Forero in 2016. In this block technique, a local anesthetic is given to the plane between the erector spinae muscle and the vertebral transverse process. The dorsal and ventral branches of the spinal nerves are blocked in this plane. However, due to individual regional anatomical differences, there is not enough data to determine the optimum volume at which the appropriate spread of local anesthetic will occur. Volume-based cadaver studies have some handicaps since they do not have the characteristics of living tissue.

This study aims to compare the postoperative analgesic efficacy of ESP block applied at the same dose but with different local anesthetic volumes in cardiac surgeries to be performed with sternotomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who will undergo coronary artery bypass grafting surgery with median sternotomy

Exclusion Criteria:

* Emergency surgeries
* Patients with allergic reactions to anesthesia and analgesia drugs to be used
* Patients who do not want to participate in the study voluntarily
* Severe systemic disease (kidney, liver, pulmonary, endocrine)
* Substance abuse history
* History of chronic pain
* Psychiatric problems and communication difficulties
* Patients who need revision due to hemostasis in the postoperative period
* Patients with severe hemodynamic instability due to infection, heavy bleeding, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Post-extubation 1st hour measurement | 1 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Post-extubation 1st hour measurement | 1 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of nausea and vomiting, if they have nausea or vomiting it will be recorded as nausea positive or vomiting positive, otherwise it will be recorded as negative.
Post-extubation 1st hour measurement | 1 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of rescue analgesic, when patients have more than 4 visual analog score (VAS), they will be administered 1mg/kg tramadol and it will be recorded.
Post-extubation 2nd hour measurement | 2 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Post-extubation 2nd hour measurement | 2 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of nausea and vomiting, if they have nausea or vomiting it will be recorded as nausea positive or vomiting positive, otherwise it will be recorded as negative.
Post-extubation 2nd hour measurement | 2 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of rescue analgesic, when patients have more than 4 visual analog score (VAS), they will be administered 1mg/kg tramadol and it will be recorded.
Post-extubation 4th hour measurement | 4 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Post-extubation 4th hour measurement | 4 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of nausea and vomiting, if they have nausea or vomiting it will be recorded as nausea positive or vomiting positive, otherwise it will be recorded as negative.
Post-extubation 4th hour measurement | 4 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of rescue analgesic, when patients have more than 4 visual analog score (VAS), they will be administered 1mg/kg tramadol and it will be recorded.
Post-extubation 8th hour measurement | 8 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Post-extubation 8th hour measurement | 8 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of nausea and vomiting, if they have nausea or vomiting it will be recorded as nausea positive or vomiting positive, otherwise it will be recorded as negative.
Post-extubation 8th hour measurement | 8 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of rescue analgesic, when patients have more than 4 visual analog score (VAS), they will be administered 1mg/kg tramadol and it will be recorded.
Post-extubation 12th hour measurement | 12 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Post-extubation 12th hour measurement | 12 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of nausea and vomiting, if they have nausea or vomiting it will be recorded as nausea positive or vomiting positive, otherwise it will be recorded as negative.
Post-extubation 12th hour measurement | 12 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of rescue analgesic, when patients have more than 4 visual analog score (VAS), they will be administered 1mg/kg tramadol and it will be recorded.
Post-extubation 24th hour measurement | 24 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Post-extubation 24th hour measurement | 24 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of nausea and vomiting, if they have nausea or vomiting it will be recorded as nausea positive or vomiting positive, otherwise it will be recorded as negative.
Post-extubation 24th hour measurement | 24 hour after endotracheal extubation, an average of 5 minutes
  patients will be evaluated in terms of rescue analgesic, when patients have more than 4 visual analog score (VAS), they will be administered 1mg/kg tramadol and it will be recorded.

SECONDARY OUTCOMES:
Mechanical ventilation duration | postoperative, approximately 4 to 10 hours
  The total time until patients suitable for endotracheal extubation
intensive care unit duration | postoperative, approximately 12 to 36 hours
  The total time until patients suitable for discharge from intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: ZELİHA A DEMİR, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Select State/Province, Turkey (Türkiye)

REFERENCES:
- [Background] Mueller XM, Tinguely F, Tevaearai HT, Revelly JP, Chiolero R, von Segesser LK. Pain location, distribution, and intensity after cardiac surgery. Chest. 2000 Aug;118(2):391-6. doi: 10.1378/chest.118.2.391. PMID 10936130
- [Background] Milgrom LB, Brooks JA, Qi R, Bunnell K, Wuestfeld S, Beckman D. Pain levels experienced with activities after cardiac surgery. Am J Crit Care. 2004 Mar;13(2):116-25. PMID 15043239
- [Background] Cheng DC, Wall C, Djaiani G, Peragallo RA, Carroll J, Li C, Naylor D. Randomized assessment of resource use in fast-track cardiac surgery 1-year after hospital discharge. Anesthesiology. 2003 Mar;98(3):651-7. doi: 10.1097/00000542-200303000-00013. PMID 12606909
- [Background] Silbert BS, Santamaria JD, Kelly WJ, O'brien JL, Blyth CM, Wong MY, Allen NB; Fast Track Cardiac Care Team. Early extubation after cardiac surgery: emotional status in the early postoperative period. J Cardiothorac Vasc Anesth. 2001 Aug;15(4):439-44. doi: 10.1053/jcan.2001.24978. PMID 11505346
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016